CLINICAL TRIAL: NCT00269737
Title: Efficacy of TTS Fentanyl in the Management of Pain in Patients With Malignancy - Study III
Brief Title: Efficacy of the Fentanyl Transdermal Therapeutic System (TTS) in the Management of Pain in Patients With Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005980
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Pain; Cancer
Keywords: fentanyl; pain; Cancer; patch
MeSH Terms: conditions — Pain; Neoplasms

INTERVENTIONS:
Drug: Fentanyl Transdermal Therapeutic System (TTS)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of continuous use of TTS fentanyl (a transdermal patch delivering the narcotic pain reliever fentanyl) for the treatment of chronic cancer pain.

DETAILED DESCRIPTION:
Moderate to severe pain is experienced by about one-third of cancer patients during the intermediate stage of their disease. Currently used medications for the treatment of moderate to severe pain due to cancer often provide inadequate pain relief and require repeated oral administration of a narcotic. Providing prolonged, safe and effective pain relief on a continuous basis would be a major therapeutic advance in the management of cancer pain. This is an open-label pilot study to evaluate the safety and effectiveness of the fentanyl Transdermal Therapeutic System (TTS) in the management of chronic pain in patients with cancer. The initial dose of the fentanyl transdermal patch is calculated based upon the equi-analgesic potency ratio of the narcotic used prior to study entry. Four dosage strengths of the fentanyl transdermal patch are available as study medication, with a nominal delivery rate of 100, 75, 50 and 25 micrograms of fentanyl per hour. Multiple transdermal patches are worn when higher doses are required. Morphine sulfate is available as needed as rescue medication to treat breakthrough pain. After the initial application, the dose is titrated for each patient within a hospital setting over the course of 3 days, or as long as is necessary to achieve adequate pain control. Changes in dose during titration occur no more frequently than once every 24 hours. After an appropriate dose is reached, the transdermal patch is replaced every 72 hours with a new transdermal patch, applied to a fresh skin site. When discharged, patients enter a 3-week program of twice weekly nursing visits to monitor patient progress. Patients are evaluated at designated time intervals for pain intensity, vital signs, and serum fentanyl concentration. Records are kept of all concomitant medications administered during the study and any adverse events. After completion of the 3-week program, patients are given the opportunity to remain on the fentanyl Transdermal Therapeutic System (TTS) for long-term treatment of their chronic pain.

The TTS (fentanyl) transdermal patch starting dose is calculated based upon the equi-analgesic potency ratio of the narcotic used prior to study entry, titrated as needed to achieve adequate pain control. The patch is replaced every 72 hours. The treatment phase is 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of intermediate stage of malignancy, operationally defined as non-localized or metastatic disease causing moderate to severe pain
* Having a diagnosis of terminal disease, defined as life expectancy of six months or less, with moderate to severe pain associated with malignancy
* Requiring treatment with a narcotic analgesic for relief of cancer pain
* Having normal liver, kidney, and lung function, as determined by liver function tests, BUN, creatinine, and blood gases

Exclusion Criteria:

* Patients with a history of allergic reaction to narcotics
* Having a history of narcotic abuse prior to cancer diagnosis
* Unable to communicate adequately to provide information assessing the effectiveness of treatment
* Having active skin disease which precludes application of the transdermal system
* Having a history of carbon dioxide (CO2) retention or respiratory problems and who, in the physician's judgment, should not use narcotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7
Dates: Start 1986-05; Study Completion 1988-02

PRIMARY OUTCOMES:
Pain intensity at designated time intervals

SECONDARY OUTCOMES:
Pharmacokinetics; Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — Alza Corporation, DE, USA

REFERENCES:
- See also: Efficacy of TTS (fentanyl) in the management of pain in patients with malignancy Study 3 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=99&filename=CR005980_CSR.pdf